CLINICAL TRIAL: NCT03861988
Title: Double-blind Trial of Intraoperative Ketamine Versus Saline in Depressed Patients Undergoing Anesthesia for Non-cardiac Surgery
Brief Title: Intraoperative Ketamine Versus Saline in Depressed Patients Undergoing Anesthesia for Non-cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Boris D. Heifets, Assistant Professor of Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49114
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder; Surgery; Orthopedic Disorder
Keywords: depression; ketamine; anesthesia; total joint arthroplasty
MeSH Terms: conditions — Depressive Disorder, Major; Musculoskeletal Diseases; Depression | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking is for double blind phase only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Open label ketamine (Experimental): Patients will receive an intravenous ketamine infusion during surgery.
  Interventions: Drug: Ketamine
- Double blind ketamine (Experimental): Patients will receive an intravenous ketamine infusion during surgery.
  Interventions: Drug: Ketamine
- Double blind placebo (Placebo Comparator): Participants will receive placebo (normal saline infusion) during surgery.
  Interventions: Drug: Normal saline (placebo)

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg over 40 minutes, intravenous.
  Other Names: Ketalar.
  Arms: Double blind ketamine; Open label ketamine
Drug: Normal saline (placebo) — Normal saline infusion over 40 minutes, equivalent volume to ketamine infusion.
  Arms: Double blind placebo

SUMMARY:
This study evaluates whether ketamine, given as part of an anesthetic, improves depression symptoms in depressed patients undergoing non-cardiac surgery. Half of participants will receive a ketamine infusion during surgery, while the other half will receive a placebo (normal saline) during surgery.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is widely prevalent among patients preparing to have surgery, and is a known risk factor for complications after surgery, including wound infection, myocardial infarction and opioid use disorder. Ketamine has emerged as an effective, rapid-acting antidepressant therapy for patients with MDD, and may be a useful tool to prevent MDD-related morbidity in the perioperative period. Ketamine has been well studied for MDD in outpatient clinics where it is given as an infusion (0.5 mg/kg over 40 minutes) in awake patients. Ketamine is often used as part of an anesthetic cocktail in sedated or anesthetized patients, but it is unknown whether ketamine has an antidepressant effect in this context. The investigators will determine whether a ketamine infusion, compared to placebo (normal saline infusion), has an antidepressant effect when given during surgical anesthesia. If ketamine is an effective antidepressant in this population under anesthesia, its use could be incorporated into a set of interventions to minimize the perioperative complications associated with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for non-cardiac, non-intracranial surgery
* Major Depressive Disorder

Exclusion Criteria:

* Pregnant of breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris D Heifets, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Derived] Lii TR, Smith AE, Flohr JR, Okada RL, Nyongesa CA, Cianfichi LJ, Hack LM, Schatzberg AF, Heifets BD. Randomized trial of ketamine masked by surgical anesthesia in patients with depression. Nat Ment Health. 2023 Nov;1(11):876-886. doi: 10.1038/s44220-023-00140-x. Epub 2023 Oct 19. PMID 38188539
- [Derived] Lii TR, Smith AE, Flohr JR, Okada RL, Nyongesa CA, Cianfichi LJ, Hack LM, Schatzberg AF, Heifets BD. Randomized Trial of Ketamine Masked by Surgical Anesthesia in Depressed Patients. medRxiv [Preprint]. 2023 Jun 15:2023.04.28.23289210. doi: 10.1101/2023.04.28.23289210. PMID 37205558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the open-label arm, recruitment occurred between August 2019 and March 2020. For the double-blind arms, recruitment occurred between February 2020 and August 2022. In all arms, recruitment occurred in medical clinics and by telephone and video visits.
Pre-assignment Details: Five participants were recruited for an open label study to evaluate and optimize study procedures prior to randomizing participants enrolled in the double-blind trial ("Double blind ketamine" vs "Double blind placebo").
Groups:
- Open Label Ketamine; Double Blind Ketamine: Patients received intravenous ketamine (0.5 mg/kg over 40 minutes) infusion during surgery.
- Double Blind Placebo: Participants received placebo (normal saline infusion over 40 minutes) during surgery.
Period: Overall Study
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Started | 5 | 20 | 20
Completed | 5 | 19 | 19
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo | Total
Number analyzed (Participants) | 5 | 20 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.4) | 50.5 (12.0) | 51.9 (18.9) | 52.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 16 | 31
  Male | 2 | 8 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 18 | 17 | 39
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 2 | 2 | 4
  White | 5 | 13 | 13 | 31
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 20 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a 10-item scale for the evaluation of depressive symptoms (Montgomery et al 1979). Each MADRS item is rated on a 0 to 6 scale. Total score range from 0-60, where lower MADRS scores indicate lower levels of depressive symptoms. The assessment for this outcome will be taken once daily on days 1, 2 and 3 post procedure. A mixed model for repeated measures (MMRM) was used to analyze the difference in postoperative MADRS score between ketamine and placebo groups..
Time Frame: Post-intervention days 1, 2 and 3
Population: Missing data occurred when the number of participants analyzed on specific days was fewer than the overall number of participants analyzed. This situation arose when some participants did not complete the instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
score on a scale
  Day 1: number analyzed (Participants) | 5 | 20 | 19
  Day 1 | 17.0 (13.0) | 12.7 (7.6) | 16.4 (17.5)
  Day 2: number analyzed (Participants) | 5 | 20 | 19
  Day 2 | 25.4 (17.3) | 15.1 (11.1) | 17.5 (11.5)
  Day 3: number analyzed (Participants) | 4 | 19 | 20
  Day 3 | 10.5 (7.1) | 17.0 (10.5) | 17.2 (12.0)
Statistical Analysis 1: Comparison: Double Blind Ketamine vs Double Blind Placebo; Test type: Superiority; p = 0.13, Mixed Models Analysis

2. Secondary Outcome: Number of Participants With Clinical Response
Description: Clinical response defined as >=50% reduction in MADRS score from baseline. MADRS score range: 0 to 60, a lower score indicates lower severity of symptoms.
Time Frame: Post-intervention days 1, 2 and 3
Population: Includes all participants still enrolled in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
Participants
  Day 1 | 2 | 12 | 10
  Day 2 | 1 | 10 | 12
  Day 3 | 3 | 9 | 10

3. Secondary Outcome: Number of Participants With Remission
Description: Remission defined as a MADRS score of <=12 on day 14. MADRS score range: 0 to 60, a lower score indicates lower severity of symptoms.
Time Frame: Post-intervention day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 19 | 19
Participants | 3 | 8 | 10

4. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Scale Score
Description: This outcome measures self-reported symptoms of anxiety and depression on a scale that ranges from 0 to 42. A lower score indicates lower severity of symptoms.
Time Frame: Post-intervention days 1, 2, 3, 5, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
score on a scale
  Day 1: number analyzed (Participants) | 5 | 20 | 19
  Day 1 | 14.8 (8.4) | 17.8 (6.6) | 19.9 (5.5)
  Day 2: number analyzed (Participants) | 5 | 18 | 20
  Day 2 | 22.6 (12.7) | 18.8 (7.5) | 21.2 (5.9)
  Day 3: number analyzed (Participants) | 5 | 19 | 20
  Day 3 | 13.0 (9.2) | 19.3 (6.3) | 20.8 (5.4)
  Day 5: number analyzed (Participants) | 5 | 19 | 19
  Day 5 | 16.6 (10.2) | 18.3 (4.8) | 18.9 (7.3)
  Day 7: number analyzed (Participants) | 5 | 16 | 19
  Day 7 | 19.2 (10.0) | 18.4 (5.3) | 19.6 (8.1)
  Day 14: number analyzed (Participants) | 5 | 19 | 19
  Day 14 | 14.0 (9.7) | 16.4 (7.2) | 17.2 (8.5)

5. Secondary Outcome: Cumulative Opioid Use
Description: This outcome measures how many cumulative morphine-equivalents milligrams of opioid pain medication the patient has taken as an inpatient and after discharge from hospital
Time Frame: Post-intervention days 1, 2, 3, 5, 7 and 14
Population: In the open-label group, total opioid consumption was recorded only for the first 3 postoperative days
Measure: Mean (Standard Deviation); unit: milligram morphine equivalents
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
milligram morphine equivalents
  Day 1 | 108.5 (72.2) | 60.9 (60.3) | 56.1 (61.5)
  Day 2 | 249.3 (173.2) | 104.6 (109.0) | 107.7 (126.3)
  Day 3 | 361.5 (237.3) | 137.9 (165.9) | 144.3 (188.4)
  Day 5: number analyzed (Participants) | 0 | 19 | 19
  Day 5 |  | 150.6 (204.3) | 156.2 (218.7)
  Day 7: number analyzed (Participants) | 0 | 19 | 19
  Day 7 |  | 171.6 (219.0) | 163.3 (221.4)
  Day 14: number analyzed (Participants) | 0 | 19 | 19
  Day 14 |  | 206.1 (270.1) | 186.4 (242.3)

6. Secondary Outcome: Hospital Length of Stay
Description: Number of days from admission (day of surgery) through discharge after surgery.
Time Frame: Average approximately 3 days post-intervention
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
days | 3.7 (0.9) | 1.9 (1.7) | 4.0 (3.3)

7. Secondary Outcome: Brief Pain Inventory Pain Intensity Scale Score
Description: Average pain intensity in the past 24 hours, rated on a numerical scale from 0 to 10 (with 0 representing "No pain" and 10 representing "Pain as bad as you can imagine").
Time Frame: Post-intervention days 1, 2, 3, 5, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
score on a scale
  Day 1: number analyzed (Participants) | 5 | 20 | 18
  Day 1 | 4.6 (1.8) | 6.0 (2.0) | 5.2 (2.8)
  Day 2: number analyzed (Participants) | 4 | 19 | 19
  Day 2 | 5.5 (2.5) | 5.3 (2.1) | 6.0 (2.3)
  Day 3: number analyzed (Participants) | 4 | 19 | 20
  Day 3 | 3.5 (3.0) | 5.5 (1.9) | 5.2 (2.4)
  Day 5: number analyzed (Participants) | 5 | 19 | 19
  Day 5 | 4.4 (2.3) | 5.5 (1.7) | 4.4 (2.3)
  Day 7: number analyzed (Participants) | 5 | 16 | 19
  Day 7 | 4.8 (2.4) | 5.1 (2.2) | 4.4 (2.4)
  Day 14: number analyzed (Participants) | 5 | 19 | 19
  Day 14 | 4.4 (3.0) | 4.8 (1.5) | 3.7 (2.0)

8. Secondary Outcome: Brief Pain Inventory Pain Interference Scale Score
Description: Pain interference in the past 24 hours, rated on a numerical scale from 0 to 10 (with 0 representing "Does not interfere" and 10 representing "Completely interferes").
Time Frame: Post-intervention days 1, 2, 3, 5, 7 and 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
Number analyzed (Participants) | 5 | 20 | 20
units on a scale
  Day 1 | 6.0 (2.7) | 8.1 (2.6) | 7.6 (3.2)
  Day 2: number analyzed (Participants) | 4 | 19 | 19
  Day 2 | 6.3 (3.0) | 8.0 (2.5) | 8.1 (2.1)
  Day 3: number analyzed (Participants) | 4 | 20 | 20
  Day 3 | 4.8 (2.2) | 7.5 (2.6) | 7.7 (2.8)
  Day 5: number analyzed (Participants) | 5 | 19 | 19
  Day 5 | 6.6 (4.3) | 7.0 (3.0) | 7.0 (2.9)
  Day 7: number analyzed (Participants) | 5 | 17 | 17
  Day 7 | 7.6 (3.8) | 6.7 (2.8) | 7.2 (3.1)
  Day 14: number analyzed (Participants) | 5 | 19 | 19
  Day 14 | 4.8 (3.1) | 6.2 (2.2) | 5.7 (3.5)

ADVERSE EVENTS:
Time Frame: Average approximately 19 days
Description: Patients reported adverse events during follow-up assessments
Arm/Group | Open Label Ketamine | Double Blind Ketamine | Double Blind Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/20 | 2/20
Other Adverse Events (participants affected / at risk) | 1/5 | 7/20 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Ketamine (N=5) | Double Blind Ketamine (N=20) | Double Blind Placebo (N=20)
Acute pulmonary embolism (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Ketamine (N=5) | Double Blind Ketamine (N=20) | Double Blind Placebo (N=20)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Uncontrolled muscle movement in fingers (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
IV site pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical revision of implanted neurostimulator (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative delirium (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03861988/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT03861988/SAP_001.pdf